CLINICAL TRIAL: NCT00361595
Title: Open Label Proof of Concept Study of IV Zoledronic Acid (ZA) 5 mg After Forteo in Postmenopausal Women
Brief Title: Intervenous (IV) Zoledronic Acid After Forteo in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Chad Deal, M.D., Chad Deal, M.D., The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446HUS120
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2011-01-14 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Osteoporosis
Keywords: osteoporosis; zoledronic acid; forteo
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental): 5 mg zoledronic acid in a single 15 minute IV
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — 5 mg zoledronic acid administered in a single 15 minute IV
  Other Names: zometa

SUMMARY:
The purpose of this study is to evaluate the adequacy of zoledronic acid in maintaining bone mass after two years of treatment with Forteo, in postmenopausal women.

DETAILED DESCRIPTION:
This will be a single center open label proof of concept study, recruiting subjects previously treated with Forteo for at least 12 months.

A screening period of 3 to 6 weeks will precede the treatment period. At the baseline visit, patients whose eligibility is confirmed will be treated with ZA and followed for 12 months. Safety and efficacy will be assessed at regular intervals (day one, day 10, month 2, month 6, month 9 and month 12). Renal safety will be assessed prior to the i.v. dose of study medication, day 10 after the i.v. dose of study medication and at 12 months. Bone density at the lumbar spine (L1-4) and total hip will be performed at 6 months and at the end of the 12 month treatment period. Biomarker analyses for secondary endpoint will be performed for at day 10, month 2, month 6, month 9 and month 12.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women to age 85, inclusive
* Finish treatment of 12 months or longer with Forteo
* Signed informed consent prior to initiation of any study-mandated procedure.

Exclusion Criteria:

* Hip and spine DXA T-score >-1.0
* Patients with 25-(OH) vitamin D levels less than 15 ng/mL at Visit 1. (Patient can be repleted with vitamin D 50,000 units biweekly for up to 2 months and re-screened anytime during the 2 months while continuing Forteo.)
* Baseline renal insufficiency (calculated creatinine clearance less than 40.0 mL/min (MDRD) at Visit 1 and/or Visit 2 or urine dipstick greater than or equal to 2+ protein without evidence of contamination or bacteriuria (may be repeated one time at least a week apart if there is suspicion of contamination). Patients with calculated creatinine clearance equal to or greater than 40.0 mL/min and less than 60.0 mL/min or serum creatinine greater than the upper limit of normal at Visit 1 must be retested between Visit 1 and 2. Patients with calculated creatinine clearance greater than 60.0 mL/min and serum creatinine within normal limits at Visit 1 do not require re-test.
* Patients who require re-test of creatinine clearance between Visit 1 and 2 will be excluded if there is an increase in serum creatinine greater than 0.5 mg/dL between Visit 1 and Visit 2.
* Serum calcium <8.5 or >11.0 mg/dl at Visit 1
* AST or ALT greater than twice the upper limit of normal
* Serum alkaline phosphatase greater than 1.5 times the upper limit of normal (liver fraction)
* No history of retinopathy or nephropathy especially in the presence of uncontrollable IDDM with Hb1 AC > 10%
* Hypersensitivity to bisphosphonates
* Treatment with biphosphonates while on Forteo
* Prior treatment with i.v. biphosphonates
* Estrogen, calcitonin, raloxifene use prior to Forteo treatment are not exclusions, but concomitant therapy during with any bone agents during the trial will not be permitted
* Any prior use of strontium ranelate or sodium fluoride
* Chronic use of systemic corticosteroids (oral or i.v.) within the last year:

NOTE: Use of corticosteroids in forms such as topical creams, nasal or inhaled formulations or those injected locally (intra-articularly) are NOT exclusionary.

* Prior exposure to anabolic steroids or growth hormone within 6 months prior to randomization
* Treatment with any investigational drug(s) and/or devices within 30 days prior to randomization.
* History of iritis or uveitis, except when secondary to trauma, and must have resolved for more than 2 years prior to randomization.
* Cancer exclusions:

  * Patients with a new diagnosis or active treatment for any malignancy less than or equal to 12 months prior to Visit 1.
  * Patients with evidence of any metastases on or prior to randomization, or with a history of metastases
  * Subjects with evidence of paraneoplastic syndrome, especially those characterized by hypercalcemia during screening or by history
  * Patients with the following may be included: basal cell or squamous cell carcinoma of the skin, colonic polyps with non-invasive malignancy which have been removed, and Carcinoma in-situ (CIS) of the prostate (Stage I only) that has been surgically removed.
* Previous major solid organ or bone marrow transplant recipient or on a transplant waiting list
* Any disease of the spine that would preclude the proper acquisition of a lumbar spine DXA (L1-L4) e.g., implantable devices, scoliosis, ankylosing spondylitis, DJD. (Less than two lumbar spine vertebral bodies evaluable)
* Active primary hyperparathyroidism or hypoparathyroidism
* Subject with complete thyroidectomy
* Active hyperthyroidism
* Hypothyroidism not treated with adequate replacement therapy
* History of multiple myeloma or Paget's disease
* Patients with severe dental problems or current dental infections, or with recent or impending dental surgery within three months of dosing
* Any medical or psychiatric condition which, in the opinion of the investigator, would preclude the participant from adhering to the protocol or completing the trial per protocol

Max Age: 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Deal, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment, 35 Subjects Start date: August, 2006 Completion date: April, 2008 Study took place at an academic medical center, recruiting subjects from investigator's practice.
Groups:
- Open Label: 5 mg zoledronic acid in a single 15 minute IV (intervenous)
Period: Overall Study
Arm/Group | Open Label
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Spine BMD (Bone Mineral Density) in g/cm^2 From Baseline to Month 12 Relative to Baseline as Measured by DXA (Dual-energy X-ray Absorptiometry)
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | Open Label
Number analyzed (Participants) | 35
grams/cm^2 | 2.2 (.036)

2. Secondary Outcome: Change in Bone Density (Grams/cm^2) at the Total Hip at 6 and 12 Months
Description: Change in bone density (grams/cm^2) at the total hip at 6 and 12 months. 12 month reported based on usual interval for bone density follow-up in clinical practice.
Time Frame: 6 months and 12 months
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | Open Label
Number analyzed (Participants) | 35
grams/cm^2 | 2.4 (.031)

3. Secondary Outcome: Change in Serum C-telopeptide Type 1 Collagen (CTX) (at Day 10 and Months 2, 6, 9 and 12)
Description: Change in serum c-telopeptide type 1 collagen (CTX) (at day 10 and months 2, 6, 9 and 12. 12 month values reported based on 12 month duraton of zolendronic acid effect.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Open Label
Number analyzed (Participants) | 35
ng/ml | -49.1 (37.6)

4. Secondary Outcome: Change in Serum N-propeptide Type 1 Collagen (P1NP) (at Day 10 and Months 2, 6, 9 and 12)
Description: Change in serum n-propeptide type 1 collagen (P1NP) (at day 10 and months 2, 6, 9 and 12. 12 month values reported based on 12 month duraton of zolendronic acid effect.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Open Label
Number analyzed (Participants) | 35
mcg/ml | -66.2 (29.1)

ADVERSE EVENTS:
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 8/35
OTHER ADVERSE EVENTS (reported when occurring in more than 3.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=35)
Transient increase in serum creatinine (Blood and lymphatic system disorders) | 2 (2)
Flu-like symptoms (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No